CLINICAL TRIAL: NCT03352154
Title: Long Latency Auditory Evoked Potentials (P300) Outcomes in Patients With Unilateral Cochlear Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Apoio ao Ensino, Pesquisa e Assistência do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (Other)
Responsible Party: Principal Investigator, Miguel Angelo Hyppolito, Head of Otolaryngology, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38224814.2.0000.5440
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Hearing Loss, Sensorineural; Deafness
Keywords: cochlear implant; Evoked Potential P300
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness

STUDY DESIGN:
Intervention Model Description: Verify the alteration of the latency and amplitude of the P300 as markers of the cognitive response after Cochlear Implant Assist in prognosis after implantation cochlear implant.
Masking Description: Not Apply
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with unilateral cochlear implants submitted to P300 (Experimental): Patients with unilateral cochlear implants, using the speech processor at least 6 months, submitted to P300 exam before CI surgery, on speech processor activation and after 06 months.
  Interventions: Diagnostic Test: P300 - Auditory long latency potential

INTERVENTIONS:
Diagnostic Test: P300 - Auditory long latency potential — Perform the P300 exams.

SUMMARY:
Bilateral severe to profound hearing loss is a socially disabling handicap. Cochlear implants can be used to improve hearing in cases where conventional hearing aids are not effective. There are few studies about the long latency Auditory Evoked Potential (P300), in individuals with hearing loss and Cochlear Implant (CI) users. The aim of this project is to study the behavior of P300 in users of unilateral CI.

DETAILED DESCRIPTION:
Bilateral severe to profound hearing loss is a socially disabling handicap. Cochlear implants can be used to improve hearing in cases where conventional hearing aids are not effective. There are few studies about the long latency Auditory Evoked Potential (P300), in individuals with hearing loss and Cochlear Implant (CI) users. The aim of this project is to study the behavior of P300 in users of unilateral CI. Twenty patients with bilateral severe and/or profound post-lingual deafness, all submitted to CI surgery, will be evaluated. Patients will be evaluated through P300 testing on the day before CI surgery, on the day of device activation and 6 months after device use. It is hoped that this study can contribute to the understanding of the mechanisms of brain plasticity involved in the recovery of hearing function after CI surgery. There are few studies on the behavior of P300 in CI users and there are no studies showing how central stimulation occurs after device implantation, during the phases of pre CI, CI activation and 6 months after CI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-lingual hearing loss undergoing cochlear implant surgery

Exclusion Criteria:

* Prelingual hearing loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2016-11-20 (Actual); Primary Completion 2020-06-04 (Estimated); Study Completion 2020-06-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of the P300 Responses after CI | 06 months after CI
  Improving the cognitive process on CI receivers

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Hyppolito, MD/PhD, Study Chair — Coordinator Health Auditory Care Program of the HCRP-FMRP-USP

IPD SHARING:
Plan to Share IPD: Yes
Include researchers on the support team.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years
Access Criteria: Free to all IPD.

REFERENCES:
- [Background] McPherson, D.L. Late potentials of the auditory system. San Diego: Singular Publishing Group; 1996.
- [Background] Groenen PA, Makhdoum M, van den Brink JL, Stollman MH, Snik AF, van den Broek P. The relation between electric auditory brain stem and cognitive responses and speech perception in cochlear implant users. Acta Otolaryngol. 1996 Nov;116(6):785-90. doi: 10.3109/00016489609137926. PMID 8973707
- [Result] Kileny PR. Use of electrophysiologic measures in the management of children with cochlear implants: brainstem, middle latency, and cognitive (P300) responses. Am J Otol. 1991;12 Suppl:37-42; discussion 43-7. PMID 2069187
- [Result] Duarte Josilene Luciene, Alvarenga Kátia de Freitas, Costa Orozimbo Alves. Potencial cognitivo P300 realizado em campo livre: aplicabilidade do teste. Rev. Bras. Otorrinolaringol. [Internet]. 2004 Dec [cited 2015 May 02] ; 70( 6 ): 780-785.
- [Result] Micco AG, Kraus N, Koch DB, McGee TJ, Carrell TD, Sharma A, Nicol T, Wiet RJ. Speech-evoked cognitive P300 potentials in cochlear implant recipients. Am J Otol. 1995 Jul;16(4):514-20. PMID 8588653
- [Result] Jordan K, Schmidt A, Plotz K, von Specht H, Begall K, Roth N, Scheich H. Auditory event-related potentials in post- and prelingually deaf cochlear implant recipients. Am J Otol. 1997 Nov;18(6 Suppl):S116-7. PMID 9391625
- [Result] Muhler R, Ziese M, Kevanishvili Z, Schmidt M, von Specht H. Visualization of stimulation patterns in cochlear implants: application to event-related potentials (P300) in cochlear implant users. Ear Hear. 2004 Apr;25(2):186-90. doi: 10.1097/01.aud.0000120366.80555.2a. PMID 15064663
- [Result] Klem GH, Luders HO, Jasper HH, Elger C. The ten-twenty electrode system of the International Federation. The International Federation of Clinical Neurophysiology. Electroencephalogr Clin Neurophysiol Suppl. 1999;52:3-6. No abstract available. PMID 10590970
- [Result] Kelly AS, Purdy SC, Thorne PR. Electrophysiological and speech perception measures of auditory processing in experienced adult cochlear implant users. Clin Neurophysiol. 2005 Jun;116(6):1235-46. doi: 10.1016/j.clinph.2005.02.011. Epub 2005 Apr 26. PMID 15978485
- [Result] Diniz Junior J, Mangabeira-Albernaz PL, Munhoz MS, Fukuda Y. Cognitive potentials in children with learning disabilities. Acta Otolaryngol. 1997 Mar;117(2):211-3. doi: 10.3109/00016489709117772. PMID 9105451
- [Result] Calhau CM, Lima Junior LR, Reis AM, Capistrano AK, Lima Ddo V, Calhau AC, Rodrigues Junior Fde A. [Etiology profile of the patients implanted in the cochlear implant program]. Braz J Otorhinolaryngol. 2011 Jan-Feb;77(1):13-8. doi: 10.1590/S1808-86942011000100003. PMID 21340183
- [Result] Beynon AJ, Snik AF, Stegeman DF, van den Broek P. Discrimination of speech sound contrasts determined with behavioral tests and event-related potentials in cochlear implant recipients. J Am Acad Audiol. 2005 Jan;16(1):42-53. doi: 10.3766/jaaa.16.1.5. PMID 15715067
- [Result] Okusa M, Shiraishi T, Kubo T, Nageishi Y. Effects of discrimination difficulty on cognitive event-related brain potentials in patients with cochlear implants. Otolaryngol Head Neck Surg. 1999 Nov;121(5):610-5. doi: 10.1016/S0194-5998(99)70067-7. PMID 10547481